CLINICAL TRIAL: NCT06386575
Title: Effect of Supra-inguinal Fascia Iliaca Block on Recovery and Recovery Quality After Total Knee Arthroplasty: A Multicenter, Prospective Randomized Controlled, Double-blind Study.
Brief Title: Suprainguinal Fascia Iliaca Block in Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Muhammed Halit Satici, Specialist, Department of Anesthesiology, Konya City Hospital, M.D, Konya City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: suprainguinal
Record Dates: First submitted 2024-04-15; First posted 2024-04-26 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Analgesia; Anesthesia, Local
MeSH Terms: conditions — Agnosia | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Suprainguinal fascia iliaca block will be applied to the patients at the end of the surgery.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Other)
  Interventions: Other: control group; Patients who received physiological saline
- suprainguinal fascia iliaca block (Active Comparator)
  Interventions: Other: suprainguinal fascia block; Patients receiving local anesthetic

INTERVENTIONS:
Other: control group; Patients who received physiological saline — All patients will be given 1 gram of paracetamol intravenously + 20 milligrams of tenoxicam + 8 milligrams of decort intravenously. Paracetamol 3x1 gram + tenoxicam 2x20 milligrams will continue to be administered. Patients in the control group will be given 40 milliliters of physiological saline during the suprainguinal fascia iliaca block.
  Arms: control group
Other: suprainguinal fascia block; Patients receiving local anesthetic — All patients will be given 1 gram of paracetamol intravenously + 20 milligrams of tenoxicam + 8 milligrams of decort intravenously. Paracetamol 3x1 gram + tenoxicam 2x20 milligrams will continue to be administered. Patients in the sfıb group will be given 40 milliliters of 0.25 % bupivacaine during the suprainguinal fascia iliaca block.
  Arms: suprainguinal fascia iliaca block

SUMMARY:
Total knee arthroplasty is the most commonly performed orthopedic surgery, especially in patients with advanced gonarthrosis and limited joint movement. After total knee arthroplasty, patients experience unbearably severe pain. Pain that is not adequately treated in the postoperative period increases the stress response in patients, increases the risk of embolism, causes bleeding in the surgical area, and causes undesirable conditions such as agitation and delirium in patients. This postoperative pain is successfully treated with various variants of multimodal analgesia.

DETAILED DESCRIPTION:
Total knee arthroplasty is the most commonly performed orthopedic surgery, especially in patients with advanced gonarthrosis and limited joint movement. After total knee arthroplasty, patients experience unbearably severe pain. Pain that is not adequately treated in the postoperative period increases the stress response in patients, increases the risk of embolism, causes bleeding in the surgical area, and causes undesirable conditions such as agitation and delirium in patients. This postoperative pain is successfully treated with various variants of multimodal analgesia.

The primary purpose of this study is; To evaluate the effects of suprainguinal fascia iliaca block on recovery and recovery in the postoperative period in patients who will undergo total knee arthroplasty surgery, using the quality of recovery-15T score.

Secondary purpose; Postoperative rest and movement numeric rating scale, patient likert scale, first rescue analgesia duration, number of patients needing rescue analgesia, total amount of rescue analgesic consumed, complications such as nausea and vomiting, and antiemetic requirements in patients who will undergo total knee arthroplasty surgery with suprainguinal fascia iliaca block is to evaluate.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo unilateral total knee arthroplasty
* Patients who will undergo spinal anesthesia
* Patients aged 18-65 years, ASA I-III
* Patients who will stay in the hospital for at least 24 hours

Exclusion Criteria:

* Patients who do not want to give consent
* Patients who do not want spinal anesthesia
* Patients for whom regional anesthesia is contraindicated
* Patients with confusion
* Patients with coagulopathy
* Patients using anticoagulants
* Patients with infection in the area to be treated
* Those who are allergic to local anesthesia
* Emergency cases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-06-06 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-03 (Actual)

PRIMARY OUTCOMES:
quality of recovery-15T | One day
  Quality of recovery-15T scores, which show the quality of recovery of the patients, will be recorded at the 24th hour after the surgery. Quality of recovery-15T (0-150, 0= lowest degree of satisfaction, 150= highest degree of satisfaction).

CONTACTS AND LOCATIONS:
Locations (1):
- Konya City Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No